CLINICAL TRIAL: NCT02057718
Title: Open Label Study of the Efficacy and Long Term Safety of LUM001 (Maralixibat), an Apical Sodium-Dependent Bile Acid Transporter Inhibitor (ASBTi), in the Treatment of Cholestatic Liver Disease in Pediatric Patients With Progressive Familial Intrahepatic Cholestasis
Brief Title: Open Label Study to Evaluate Efficacy and Long Term Safety of LUM001 (Maralixibat) in the Treatment of Cholestatic Liver Disease in Patients With Progressive Familial Intrahepatic Cholestasis
Acronym: INDIGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM001-501; 2013-003833-14 (EudraCT Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Progressive Familial Intrahepatic Cholestasis (PFIC)
Keywords: Bile duct diseases; Intrahepatic Cholestasis; Cholestasis; PFIC; Pruritus; Cholestatic Liver Disease
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Bile Duct Diseases; Cholestasis, Intrahepatic; Cholestasis; Pruritus | interventions — maralixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM001 (Maralixibat) (Experimental): Participants will receive LUM001, also known as Maralixibat (MRX) twice a day (BID).
  Interventions: Drug: LUM001 (Maralixibat)

INTERVENTIONS:
Drug: LUM001 (Maralixibat) — LUM001 also known as Maralixibat (MRX) oral dose up to twice a day (BID).

SUMMARY:
This is an open label study in children with Progressive Familial Intrahepatic Cholestasis (PFIC) designed to evaluate the safety and efficacy of LUM001, also known as Maralixibat (MRX). Efficacy will be assessed by evaluating the effect of LUM001 on pruritus and the biochemical markers of pruritus associated with PFIC.

DETAILED DESCRIPTION:
The study is divided into 5 parts: a 4-week dose escalation period, a 4-week stable dosing period, a 5-week stable dosing period, a 59-week long-term exposure period, and an optional follow-up treatment period for eligible participants who continue treatment with LUM001. Participants in the optional follow-up treatment period will continue to receive study drug until they are eligible to enter another LUM001 study or until LUM001 is available commercially, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects between the ages of 12 months and 18 years inclusive.

2. Diagnosis of PFIC based on:

1. Intrahepatic cholestasis manifest by total serum bile acid >3x upper limit of normal (ULN) for age and, b or c:
2. Two documented mutant alleles in ATP8B1, or ABCB11.
3. Evidence of chronic liver disease, excluding those listed in (see Section 16.3), with one or more of the following criteria:

   1. Duration of biochemical or clinical abnormalities of >6 months, or
   2. Pathologic evidence of progressive liver disease, or
   3. Sibling of known individual affected by PFIC (predicted to be chronic).

   3. GGTP <100 IU/L at screening. 4. Females of childbearing potential must have a negative urine or serum pregnancy test [β human chorionic gonadotropin (β-hCG)] during screening and a negative urine pregnancy test at the Baseline (Day 0) visit.

   5. Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial, as described in Section 8.7.1. of the protocol 6. Informed consent and assent (per IRB/EC) as appropriate. 7. Access to phone for scheduled calls from study site. 8. Caregivers and children above the age of assent must have the ability to read and understand one of the following languages: English, Spanish, US Spanish, French, German or Polish.

   9. Subjects expected to have a consistent caregiver(s) for the duration of the first 13 weeks of the study.

   10. Caregivers (and age appropriate subjects) must be willing and able to use an eDiary device as required by the study. To accommodate potential cultural restrictions within the FIC1 affected population a paper version of the ItchRO diary will be made available.

   11. Caregivers (and age appropriate subjects) using the eDiary must digitally accept the licensing agreement in the eDiary software at the outset of the study.

   12. Caregivers (and age appropriate subjects) must complete at least 10 eDiary reports (morning or evening) during each of two consecutive weeks of the screening period, prior to assignment (maximum possible reports = 14 per week). Subjects using a paper diary must complete the same number of reports within the same timeframe

   Exclusion Criteria
   1. Chronic diarrhea requiring specific intravenous fluid or nutritional intervention for the diarrhea and/or its sequelae.
   2. Surgical disruption of the enterohepatic circulation at the time at screening. Subjects who have undergone reversal of a prior surgical procedure intended to disrupt enterohepatic circulation and who and have a permanently restored flow of bile acids from the liver to the terminal ileum may be eligible for the study upon consultation with the Medical Monitor.
   3. Liver transplant.
   4. Decompensated cirrhosis [international normalized ratio (INR) > 1.5, albumin < 30 g/L, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy].
   5. ALT >15×ULN at screening.
   6. History or presence of other liver disease (see Section 16.3).
   7. History or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (e.g., inflammatory bowel disease).
   8. Liver mass on imaging.
   9. Known diagnosis of human immunodeficiency virus (HIV) infection.
   10. Cancers except for in situ carcinoma, or cancers treated at least 5 years prior to screening with no evidence of recurrence.
   11. Any female who is pregnant or lactating or who is planning to become pregnant within 20 weeks of assignment.
   12. Any known history of alcohol or substance abuse.
   13. Administration of bile acid or lipid binding resins within 30 days prior to Baseline / Day 0 and throughout the trial.
   14. Administration of sodium phenylbutyrate within 30 days prior to Baseline / Day 0 and throughout the trial.
   15. Investigational drug, biologic, or medical device within 30 days prior to screening, or 5 half-lives of the study agent, whichever is longer.
   16. History of non-adherence to medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to non-adherence with the study protocol based on Investigator judgment.
   17. Any other conditions or abnormalities which, in the opinion of the Investigator or Medical monitor, may compromise the safety of the subject, or interfere with the subject participating in or completing the study

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (10):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
- Hopital Femme Mere Enfant De Lyon, Bron, France
- The Children's Memorial Health Institute, Warsaw, Poland
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - Leeds Teaching Hospital NHS Trust, Leeds
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loomes KM, Squires RH, Kelly D, Rajwal S, Soufi N, Lachaux A, Jankowska I, Mack C, Setchell KDR, Karthikeyan P, Kennedy C, Dorenbaum A, Desai NK, Garner W, Jaecklin T, Vig P, Miethke A, Thompson RJ. Maralixibat for the treatment of PFIC: Long-term, IBAT inhibition in an open-label, Phase 2 study. Hepatol Commun. 2022 Sep;6(9):2379-2390. doi: 10.1002/hep4.1980. Epub 2022 May 4. PMID 35507739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 33 participants were enrolled at 11 sites in 4 countries (US, UK, France, Poland). Participants included 19 females and 14 males ranging from 1 to 13 years of age. Screening, treatment and safety follow-up, was approximately 76 weeks after which participants had the option of continuing in the additional follow-up treatment period up to 287 weeks.
Pre-assignment Details: A total of 37 PFIC patients were screened for the study. Four of these patients were screen failures under the original protocol. A total of 33 participants were enrolled and subsequently had genotyping performed. Of the 33 participants, 8 were PFIC1 and 25 were PFIC2. Two pairs of siblings (all with PFIC2) from 2 families were enrolled. Only a single sibling from each pair was considered for the primary analysis.
Groups:
- Progressive Familial Intrahepatic Cholestasis 1 (PFIC1): Enrolled subjects with PFIC1 subtype. All subjects received Maralixibat (LUM001; MRX).
- Progressive Familial Intrahepatic Cholestasis 2 (PFIC2) (Overall): Overall PFIC2 subtype to include PFIC2 phenotype: - non-truncating (mild to moderate phenotype with residual BSEP [liver-specific transporter] function) - truncating (severe phenotype without residual BSEP function or complete absence of BSEP). All subjects received Maralixibat (LUM001; MRX).
Period: Completed Study Treatment Through Wk. 72
Arm/Group | Progressive Familial Intrahepatic Cholestasis 1 (PFIC1) | Progressive Familial Intrahepatic Cholestasis 2 (PFIC2) (Overall)
Started | 8 | 25
Completed Study Treatment Through Week 72 | 6 | 16
Completed | 6 | 16
Not Completed | 2 | 9
Not completed — Progressive disease | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Consent withdrawn by caregiver | 1 | 1
Not completed — Consent withdrawn by subject | 0 | 1
Not completed — Liver Transplant | 0 | 1
Period: Optional Follow-up Treatment Period
Arm/Group | Progressive Familial Intrahepatic Cholestasis 1 (PFIC1) | Progressive Familial Intrahepatic Cholestasis 2 (PFIC2) (Overall)
Started | 6 | 16
Completed | 4 | 8
Not Completed | 2 | 8
Not completed — Did not consent to protocol amendment | 1 | 3
Not completed — Progressive disease | 0 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Liver Transplant | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PFIC1: Sub-group analysis of enrolled subjects with PFIC1 subtype
- PFIC2 (Overall): Sub-group analysis of overall PFIC2 subtype to include PFIC2 phenotype: - non-truncating (mild to moderate phenotype with residual BSEP [liver-specific transporter] function) - truncating (severe phenotype without residual BSEP function or complete absence of BSEP)
- Total: Total of all reporting groups
Arm/Group | PFIC1 | PFIC2 (Overall) | Total
Number analyzed (Participants) | 8 | 25 | 33
Age, Customized [Number; unit: Subjects]
  <2 years | 1 | 6 | 7
  2 to 4 years | 5 | 10 | 15
  5 to 8 years | 2 | 4 | 6
  9 to 12 years | 0 | 4 | 4
  13 to 18 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 17 | 19
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 21 | 29
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 20 | 26
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 15
  Poland | 0 | 1 | 1
  United Kingdom | 3 | 11 | 14
  France | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint (Week 13) in Fasting sBA Level
Time Frame: Baseline (Day 0) to Week 13
Measure: Mean (Full Range); unit: umol/L
Groups:
- Maralixibat: All subjects received maralixibat (MRX)
- PFIC1: Enrolled subjects with PFIC1 subtype
- PFIC2 (Overall): Overall PFIC2 subtype to include PFIC2 phenotype: - non-truncating (mild to moderate phenotype with residual BSEP [liver-specific transporter] function) - truncating (severe phenotype without residual BSEP function or complete absence of BSEP)
Arm/Group | Maralixibat | PFIC1 | PFIC2 (Overall)
Number analyzed (Participants) | 31 | 8 | 23
umol/L | -23 [-463 to 279] | 18 [-117 to 149] | -38 [-463 to 279]
Statistical Analysis 1: Comparison: PFIC1 vs PFIC2 (Overall); This analysis shows the change from baseline to Week 13 in sBA levels for the overall Modified Intent-to-treat Population. Even though a comparison of PFIC1 vs PFIC2 (overall) is noted, the results are the change from baseline for all participants and is not comparative; Test type: Other — Null hypothesis (H0): mean change from baseline to Week 13 is zero. The null hypothesis was tested for each of the 2 PFIC subgroups and overall; the change in the overall population is presented here; Mean Difference (Net) = -23.304, 95% CI 2-sided [-82.35 to 35.742], Standard Deviation 160.9748

2. Secondary Outcome: Change From Baseline to Week 13/ET in Pruritus as Measured by ItchRO(Obs)
Description: This secondary efficacy endpoint is the change from baseline to Week 13 in pruritus as measured by ItchRO(Obs) weekly average morning score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe).
Time Frame: Baseline (Day 0) to Week 13
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Maralixibat | PFIC1 | PFIC2 (Overall)
Number analyzed (Participants) | 31 | 8 | 23
scores on a scale | -0.7 (0.65) | -0.8 (0.83) | -0.7 (0.59)

3. Secondary Outcome: Change From Baseline to Week 13/ET in Pruritus as Measured by ItchRO(Pt)
Description: This secondary efficacy endpoint is the change from baseline to Week 13 in pruritus as measured by ItchRO(Pt) weekly average morning score. ItchRO scores range from 0 to 4; the higher score indicates increasing itch severity (0 = none; 4 = very severe).
Time Frame: Baseline (Day 0) to Week 13
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Maralixibat | PFIC1 | PFIC2 (Overall)
Number analyzed (Participants) | 9 | 2 | 7
scores on a scale | -0.6 (0.57) | -0.4 (0.65) | -0.7 (0.57)

4. Secondary Outcome: Change From Baseline to Week 13/ET in ALT
Time Frame: Baseline (Day 0) to Week 13
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Maralixibat | PFIC1 | PFIC2 (Overall)
Number analyzed (Participants) | 31 | 8 | 23
U/L | -9 (61.8) | -2 (29.1) | -11 (70.1)

5. Secondary Outcome: Change From Baseline to Week 13/ET in Total Bilirubin
Time Frame: Baseline (Day 0) to Week 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Maralixibat | PFIC1 | PFIC2 (Overall)
Number analyzed (Participants) | 31 | 8 | 23
mg/dL | -0.2 (1.65) | -0.8 (2.95) | -0.0 (0.9)

6. Secondary Outcome: Change From Baseline to Week 13/ET in Direct Bilirubin
Time Frame: Baseline (Day 0) to Week 13
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Maralixibat | PFIC1 | PFIC2 (Overall)
Number analyzed (Participants) | 31 | 8 | 23
mg/dL | -0.1 (1.12) | -0.3 (1.93) | -0.0 (0.72)

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (up to 287 weeks)
Description: All treatment-emergent AEs, whether observed by the Investigator, reported by the subject, subject's caregiver, from laboratory findings, or other means, were recorded on the AE eCRF and medical record. 'Occurrences' relates to the number of events; 'subjects affected' relates to the number of subjects who experienced the AE. The arms were combined to have one larger analysis population, allowing for a more robust understanding of incidence rates of AEs for patients with PFIC treated with MRX.
Groups:
- Safety Population: The safety population is defined as all subjects who were assigned and received at least one dose of the study drug. Safety analysis consists of the MITT population (Modified Intent-to-Treat [MITT]). The arms have been combined to have one larger analysis population, thus allowing for a more robust understanding of the incidence rates of AEs for patients with PFIC treated with Maralixibat.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 15/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=33)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Enteral nutrition (Surgical and medical procedures) | 1 (1)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=33)
Hypertension (Vascular disorders) | 1 (1)
Spider vein (Vascular disorders) | 1 (1)
Biliary-tract operation (Surgical and medical procedures) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (7)
Pyrexia (General disorders) | 20 (83)
Fatigue (General disorders) | 4 (4)
Influenza like illness (General disorders) | 3 (3)
Malaise (General disorders) | 3 (4)
Chest pain (General disorders) | 2 (4)
Disease progression (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Calcinosis (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Injection site discomfort (General disorders) | 1 (2)
Injection site mass (General disorders) | 1 (2)
Injection site pain (General disorders) | 1 (5)
Injection site rash (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Irritability (Psychiatric disorders) | 5 (7)
Anxiety (Psychiatric disorders) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1)
Encopresis (Psychiatric disorders) | 1 (1)
Executive dysfunction (Psychiatric disorders) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Sleep terror (Psychiatric disorders) | 1 (1)
Scrotal disorder (Reproductive system and breast disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Scratch (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2)
Ear injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio increased (Investigations) | 7 (18)
Blood bilirubin increased (Investigations) | 5 (6)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
International normalised ratio abnormal (Investigations) | 2 (4)
Vitamin E decreased (Investigations) | 2 (3)
Bilirubin conjugated increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (2)
Human rhinovirus test positive (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Protein C deficiency (Congenital, familial and genetic disorders) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (39)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (15)
Encephalopathy (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2)
Migraine (Nervous system disorders) | 1 (4)
Paraesthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (3)
Seizure (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 5 (9)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (2)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 19 (70)
Abdominal pain (Gastrointestinal disorders) | 15 (34)
Abdominal pain upper (Gastrointestinal disorders) | 8 (37)
Faeces pale (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 5 (6)
Toothache (Gastrointestinal disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 17 (38)
Frequent bowel movements (Gastrointestinal disorders) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (3)
Teething (Gastrointestinal disorders) | 2 (3)
Anal haemorrhage (Gastrointestinal disorders) | 1 (2)
Defaecation urgency (Gastrointestinal disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 2 (3)
Chromaturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (6)
Jaundice (Hepatobiliary disorders) | 3 (4)
Hepatic mass (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Ocular icterus (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (19)
Rash (Skin and subcutaneous tissue disorders) | 5 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Spider naevus (Skin and subcutaneous tissue disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Clubbing (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Delayed puberty (Endocrine disorders) | 1 (1)
Growth hormone deficiency (Endocrine disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Vitamin E deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (49)
Upper respiratory tract infection (Infections and infestations) | 11 (35)
Gastroenteritis (Infections and infestations) | 4 (4)
Varicella (Infections and infestations) | 5 (5)
Conjunctivitis (Infections and infestations) | 4 (5)
Ear infection (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 4 (7)
Viral infection (Infections and infestations) | 4 (7)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 3 (4)
Tooth abscess (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (9)
Body tinea (Infections and infestations) | 2 (2)
Epstein-Barr virus infection (Infections and infestations) | 2 (2)
Eye infection (Infections and infestations) | 2 (3)
Fungal skin infection (Infections and infestations) | 2 (3)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 2 (3)
Pharyngitis (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3)
Bronchitis (Infections and infestations) | 1 (8)
Candida infection (Infections and infestations) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Genital infection fungal (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lice infestation (Infections and infestations) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Viral pharyngitis (Infections and infestations) | 1 (1)
Ear infection viral (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analyzed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT02057718/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02057718/SAP_001.pdf